CLINICAL TRIAL: NCT02868073
Title: A Phase 1, Randomized, Double-Blind, Placebo-controlled, Dose-ranging Trial to Determine the Safety and Immunogenicity of an Adenoviral-vector Based Norovirus Vaccine (VXA-G1.1-NN) Expressing GI.1 VP1 and dsRNA Adjuvant Administered Orally to Healthy Volunteers
Brief Title: Phase 1 Placebo-controlled, Randomized Trial of an Adenoviral-vector Based Norovirus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VXA-G11-101
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Norovirus Gastroenteritis
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- H1N1 (high dose) Oral Vaccine Tablet (Experimental): Singe dose of orally administered VXA-G1.1-NN (high dose) Oral Vaccine Tablet. VXA-G1.1-NN is an E1/E3-deleted replication-defective Adenovirus serotype 5 vaccine vector for prevention of noroviral gastroenteritis caused by Norovirus GI.1. The vaccine vector encodes for a full length VP1 (major capsid protein) gene from Norvirus GI.1 Norwalk.
  Interventions: Biological: VXA-G1.1-NN (high dose) Oral Vaccine Tablet
- H1N1 (low dose) Oral Vaccine Tablet (Experimental): Singe dose of orally administered VXA-G1.1-NN (low dose) Oral Vaccine Tablet. VXA-G1.1-NN is an E1/E3-deleted replication-defective Adenovirus serotype 5 vaccine vector for prevention of noroviral gastroenteritis caused by Norovirus GI.1. The vaccine vector encodes for a full length VP1 (major capsid protein) gene from Norvirus GI.1 Norwalk.
  Interventions: Biological: VXA-G1.1-NN (low dose) Oral Vaccine Tablet
- Placebo Tablets (Placebo Comparator): Singe dose of VXA Placebo tablets. The placebo tablets are small off-white tablets that are similar in size and number to the active vaccine dose being delivered.
  Interventions: Other: VXA Placebo Tablets

INTERVENTIONS:
Biological: VXA-G1.1-NN (high dose) Oral Vaccine Tablet — The drug product will be provided as small white enteric-coated tablets. Multiple tablets will be administered to deliver the high dose.
  Other Names: H1N1 (high dose) Oral Vaccine Tablet
  Arms: H1N1 (high dose) Oral Vaccine Tablet
Other: VXA Placebo Tablets — The placebo will be provided as small white enteric-coated tablets that are similar in size and number to the active drug product tablets.
  Other Names: Placebo Control
  Arms: Placebo Tablets
Biological: VXA-G1.1-NN (low dose) Oral Vaccine Tablet — The drug product will be provided as small white enteric-coated tablets. Multiple tablets will be administered to deliver the low dose.
  Other Names: H1N1 (low dose) Oral Vaccine Tablet
  Arms: H1N1 (low dose) Oral Vaccine Tablet

SUMMARY:
A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Trial to Determine the Safety and Immunogenicity of an Adenoviral-Vector Based Norovirus Vaccine (VXA-G1.1-NN) Expressing GI.1 VP1 and dsRNA Adjuvant Administered Orally to Healthy Volunteers

DETAILED DESCRIPTION:
The study will enroll 66 subjects in four cohorts. All subjects will receive a single administration of VXA-G1.1-NN at a low dose, a high dose or placebo.

Two sentinel groups will enroll 3 subjects each in an open-label manner (Cohorts 1 and 3) to receive VXA-G1.1-NN prior to enrolling either of the randomized, controlled cohorts (Cohorts 2 and 4). Within the double-blinded Cohorts (2 and 4), placebo subjects will receive the same number of tablets as the vaccine subjects in that Cohort. Subjects will be enrolled and dosed in the low dose groups prior to initiation of dosing in the high dose group.

Cohort 1: 3 subjects at low dose Cohort 2: 20 subjects at low dose and 10 placebo Cohort 3: 3 subjects at high dose Cohort 4: 20 subjects at low dose and 10 placebo

Subjects will be followed for 28 days post vaccination for preliminary immunogenicity. Subjects will continue to be followed for 1 year post-vaccination for long term safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged 18 - 49 years, inclusive
2. Able to give written informed consent
3. Healthy (no clinically significant health concerns)
4. Safety laboratory values within the following range criteria normal range
5. Body mass index between 17 and 35 at screening

Exclusion Criteria:

1. Receipt of any investigational norovirus vaccine within two years prior to study
2. Receipt of any investigational vaccine, drug or device within 8 weeks preceding vaccination
3. Administration of any licensed vaccine within 30 days prior to study
4. Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical/surgical treatment or significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed at baseline
5. History of drug, alcohol or chemical abuse within 1 year prior to vaccination
6. Presence of a fever ≥ 38oC measured orally at baseline
7. Stool sample with occult blood at screening -

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Solicited and Unsolicited Adverse Events | Day 1 thru Day 28
  Solicited Symptoms of Reactogenicity (thru Day 8); unsolicited Adverse Events thru Day 28 post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sterling, MD, PhD, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim L, Liebowitz D, Lin K, Kasparek K, Pasetti MF, Garg SJ, Gottlieb K, Trager G, Tucker SN. Safety and immunogenicity of an oral tablet norovirus vaccine, a phase I randomized, placebo-controlled trial. JCI Insight. 2018 Jul 12;3(13):e121077. doi: 10.1172/jci.insight.121077. PMID 29997294